CLINICAL TRIAL: NCT05295147
Title: The Effect of Palmar Grasp Reflex Stimulation on Physiological Parameters and Crying Time in the Newborn Bath
Brief Title: Physiological Parameters and Crying Time in the Newborn Bath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: MSc Elif Simay KOÇ (Unknown)
Responsible Party: Principal Investigator, Türkan Kadiroğlu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/51
Record Dates: First submitted 2022-03-07; First posted 2022-03-24 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Infant, Newborn

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palmar Grasp Reflex Stimulation (Experimental)
  Interventions: Other: Palmar Grasp Reflex Stimulation
- Control Group (No Intervention)

INTERVENTIONS:
Other: Palmar Grasp Reflex Stimulation — The palmar grasp reflex is an involuntary flexion-adduction movement involving the hands and fingers.
  Arms: Palmar Grasp Reflex Stimulation

SUMMARY:
Bathing is essential for maintaining and improving the health of the newborn. It has numerous beneficial effects, such as cleaning and protecting the skin, preventing infections, cleaning unwanted substances, regulating blood circulation and the respiratory system, regulating body temperature, relieving pain, providing comfort, and supporting the parent-infant bond. Although bathing has many benefits, it is a stressful experience for newborn babies. Research on the effects of bathing on babies has shown that babies experience behavioral difficulties during bathing, such as crying, restlessness, hiccups, yawning, tremors, body looseness, looseness of the extremities, facial looseness, opening of fingers, and grimacing. Bathing may also lead to some physiological responses, such as hypothermia, hypoxia, dyspnea, cyanosis, desaturation, and tachycardia.Therefore, this study aimed to determine the effect of palmar grasp reflex stimulation during neonatal bath on the physiological parameters and crying time of the newborn.

ELIGIBILITY:
Inclusion Criteria:

* At least 24 hours after birth
* have a gestational age over 36
* not be asphyxiated
* Feeding at least 1-3 hours before bathing
* Not receiving analgesic sedation before bathing
* Stable vital signs

Exclusion Criteria:

• Ineligible for immersion tub bathing

Ages: 2 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Body temperature in Celsius | 12 week
Respiratory rate per minute | 12 week
Pulse per minute | 12 week
Oxygen saturation levels in % | 12 week
Crying time in seconds | 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- AtaturkU, Yakutiye, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No